CLINICAL TRIAL: NCT06462703
Title: Tablet-based Application for Cognitive Therapy In the Care of Brain Injury
Brief Title: Tablet-based Application for Cognitive Therapy
Acronym: TACTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Floridsdorf (Other)
Responsible Party: Principal Investigator, Peter Lackner, Prof. Dr., Klinikum Floridsdorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TACTIC
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients allocated to the intervention group receive treatment through the myReha therapy software in addition to their usual standard care (i.e., care-as-usual; CAU)
  Interventions: Device: Tablet-based neurorehabilitation with myReha
- Control Group (No Intervention): Patients allocated to the control group only receive usual standard care (CAU).

INTERVENTIONS:
Device: Tablet-based neurorehabilitation with myReha — The myReha therapy software provides cognitive therapy in the domains attention, executive functions, perception, language, speech, arithmetics, and memory. It automatically creates weekly plans that are individually tailored to a patient's abilities and provides real-time feedback when completing tasks. Intelligent algorithms ensure that the exercises always remain at the optimum level of difficulty.
  Arms: Intervention Group

SUMMARY:
Cognitive impairments such as deficits in attention, executive functions, perception, language, speech, arithmetics, and memory are very common symptoms after acquired brain injury, which can be caused by neurological diseases such as stroke, cerebral haemorrhage or traumatic brain injury. Around 83% of patients with brain injury suffer from a sequelae of cognitive impairments.

Since the effects caused by neurological diseases can vary greatly from person to person, intensive and individual neuro-rehabilitation is necessary to help patients return to an independent life in the best possible way. In the DACH area (i.e., in Germany, Austria, and Switzerland), patients with cognitive impairments following brain injuries generally receive this intensive and interdisciplinary treatment while being hospitalised in an inpatient clinic following acute medical care.

However, once they leave inpatient care facilities, there are insufficient treatment options readily available to them due to limitations/shortages in the healthcare system's resources, although studies indicate that an increase in therapy time (both in outpatient settings at home or in care facilities) enables greater, long-term rehabilitation progress and faster reintegration and participation in everyday life. Thanks to recent technical advancements, digital treatment options now promise the availability of sufficiently frequent and intensive treatment outside of clinic settings. In that context, the myReha therapy software (available as an app on iOS ad Android tablets), a certified medical device, was developed to enable patients to receive individualised and intensive therapy regardless of the healthcare system's constraints. To test the effectiveness of the myReha therapy software, in this two-arm, randomised, controlled study, patients in the intervention group receive treatment through the myReha therapy software in addition to their usual standard care (i.e., care-as-usual - CAU), while the control group only receives CAU. Treatment outcomes (i.e., rehabilitation progress) are measured based on the CERAD-plus.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive impairment (deficits in attention, arithmetics, executive functions, memory, language, perception) according to CERAD-plus after a diagnosed brain injury ≥ 4 weeks ago
* No prior experience with a therapy app for neurological deficits
* Motivation to use the therapy software regularly
* Sufficiently good German language skills prior to the brain injury

Exclusion Criteria:

* Being unable to use a tablet without assistance
* Severe visual or hearing impairment that interferes with the performance on psychometric testing procedures
* Any pre-existing speech or language disorder or dementia prior to the onset of brain injury
* An ongoing outpatient or inpatient rehabilitation at the time of study inclusion or planned rehabilitation of the primary disease during the study period
* Serious disabling disease(s) which, in the opinion of the investigator, would preclude participation in the study until the follow-up phase
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in CERAD-plus scores | From enrolment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
Mean change from baseline in BIAS-R scores | From enrolment to the end of treatment at 12 weeks
Mean change from baseline in CETI score | From enrolment to the end of treatment at 12 weeks
Mean change from baseline in HADS-D scores | From enrolment to the end of treatment at 12 weeks
Mean change from baseline in EQ-5D-5L scores | From enrolment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Floridsdorf, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No